CLINICAL TRIAL: NCT06131671
Title: Effects of Whole-body Electrostimulation on Functional Mobility and Quality of Life in the Elderly: Randomized Clinical Trial
Brief Title: Whole-body Electrostimulation on Functional Mobility and Quality of Life in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Leonhardt Ventures LLC (Industry)
Responsible Party: Principal Investigator, Jociane Schardong, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BS_Eldery
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Aged
Keywords: Aged; Electric stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive whole-body electrical stimulation associated with exercises for upper, lower limbs and trunk for twice a week, for eight weeks, totaling 16 sessions.
  Interventions: Other: Whole-body electrical stimulation
- Control (No Intervention): This group will not receive any type of electrical stimulation or exercise.

INTERVENTIONS:
Other: Whole-body electrical stimulation — The parameters adopted for the treated group will be: symmetrical biphasic current, pulse width of 400 µs, frequency of 80 Hz, contraction time of five seconds and decreasing rest time, varying from 10 to 5 s. The intensity will be individually adjusted to the patient's maximum tolerance limit to produce visible muscle contraction.
  The session time will be 15 to 20 minutes and the number of contractions will increase with each week of training.
  Concomitant to the electrical stimuli, exercises will be performed for the elbow flexors and extensors, spine flexors and extensors, knee flexors and extensors, hip flexors and extensors and the calf muscles.
  Other Names: Whole-body electromyostimulation
  Arms: Intervention

SUMMARY:
Elderly people experience reduced strength, mass and muscle function throughout the aging process, and this negatively affects the functionality and quality of life of these individuals. A randomized clinical trial will be carried out with 30 volunteers who will be allocated into two groups (whole-body electrical stimulation or control). Whole-body electrical stimulation (WBS) sessions will take place twice a week, for 8 weeks, totaling 16 sessions. The primary outcomes of this study are functional mobility (Timed Up and Go test) and quality of life (EQ-5D questionnaire). Functional mobility will be assessed at baseline, after 4 and 8 weeks of treatment or follow-up. Quality of life will be assessed only at the beginning and end of 8 weeks.

DETAILED DESCRIPTION:
Elderly people experience reduced strength, mass and muscle function throughout the aging process, and this negatively affects the functionality and quality of life of these individuals. Rehabilitation strategies similar to conventional exercise that minimize the damage caused by aging and improve subjects' adherence need to be studied. A randomized clinical trial will be carried out with 30 volunteers who will be allocated into two groups (whole-body electrical stimulation or control). Whole-body electrical stimulation (WBS) sessions will take place twice a week, for 8 weeks, totaling 16 sessions. Simultaneously with the WBS, the elderly will perform exercises for the upper, lower limbs and trunk. The following assessments will be carried out at baseline and 8 weeks to verify the effect of therapy: assessment of functional mobility; quality of life (EQ-5D); isometric muscle strength of the quadriceps muscles, biceps brachii and handgrip strength; lower limb muscle strength; assessment of body composition; assessment of cellular senescence; the inflammatory profile; well-being; measurement of muscle damage and pain; assessment of therapy safety and assessment of sleep quality. Assessments of functional mobility, lower limb muscle strength, cellular senescence; the inflammatory profile; well-being; and muscle damage will also be carried out in 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people aged between 60 and 85 years;
* Both sexes;
* To have the ability to walk.

Exclusion Criteria:

* Cognitive dysfunction;
* Intolerance to electrical stimulator and/or changes in skin sensitivity;
* Skin injuries or burns where the electrodes are positioned;
* Sequelae of stroke;
* Recent acute myocardial infarction;
* Uncontrolled hypertension;
* Grade IV heart failure or decompensated;
* Unstable angina or arrhythmia;
* Peripheral vascular changes in the lower limbs such as venous thrombosis deep;
* Disabling osteoarticular or musculoskeletal disease;
* Uncontrolled diabetes;
* Cancer;
* Autoimmune disease;
* Pacemaker;
* Epilepsy;
* Hemophilia;
* Chronic obstructive pulmonary disease;
* Liver and kidney diseases;
* Grade II obesity (BMI≥35).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Functional mobility. | Baseline, after 4 and 8 weeks.
  Functional mobility will be assessed using the "Timed Up and Go" test.
Change in quality of life measured by the EuroQol five-dimensional questionnaire (EQ-5D). | Baseline and after 8 weeks.
  Change in quality of life will be assessed by the EuroQol five-dimensional questionnaire (EQ-5D). The final score of this questionnaire can vary from 0 to 1. The closer to 1, the better the subject's quality of life.

SECONDARY OUTCOMES:
Isometric muscle strength of the quadriceps muscle. | Baseline and after 8 weeks.
  Isometric muscle strength of the quadriceps muscle will be assessed by dynamometry.
Isometric muscle strength of the biceps brachii. | Baseline and after 8 weeks.
  Isometric muscle strength of the quadriceps muscle will be assessed by dynamometry.
Isometric handgrip strength. | Baseline and after 8 weeks.
  Isometric handgrip strength will be assessed by dynamometry.
Lower limb muscle strength. | Baseline, after 4 and 8 weeks.
  Lower limb muscle strength will be assessed by the 10-repetition sit-stand test (SST10).
Body composition. | Baseline and after 8 weeks.
  Body composition will be assessed by bioimpedance.
Cellular senescence. | Baseline, after 4 and 8 weeks.
  Cellular senescence will be assessed by measuring alpha-klotho protein by ELISA.
Inflammatory profile. | Baseline, after 4 and 8 weeks.
  Inflammatory profile will be assessed by measuring interleukin 6 by ELISA.
Inflammatory profile. | Baseline, after 4 and 8 weeks.
  Inflammatory profile will be assessed by measuring interleukin 10 by ELISA.
Inflammatory profile. | Baseline, after 4 and 8 weeks.
  Inflammatory profile will be assessed by measuring tumor necrosis factor alpha by ELISA.
Well-being. | Baseline, after 4 and 8 weeks.
  Well-being will be assessed by measuring beta-endorphin by ELISA.
Muscle damage. | Baseline, after 4 and 8 weeks.
  Muscle damage will be assessed by creatine kinase dosage.
Muscle pain measured by analogic visual scale (AVS). | Baseline and after 8 weeks.
  Muscle pain will be assessed by analogic visual scale (AVS). This scale ranges from 0 to 10. The closer to 10, the greater the subject's pain.
Sleep quality. | Baseline and after 8 weeks.
  Sleep quality will be assessed by Pittsburgh Sleep Quality Index (PSQI).
Change in heart rate. | Baseline and after 20 minutes of whole-body electrical stimulation.
  Safety will be assessed by monitoring heart rate by pulse oximetry.
Change in peripheral oxygen saturation. | Baseline and after 20 minutes of whole-body electrical stimulation.
  Safety will be assessed by monitoring peripheral oxygen saturation by pulse oximetry.
Change in systolic blood pressure. | Baseline and after 20 minutes of whole-body electrical stimulation.
  Safety will be assessed by monitoring systolic blood pressure by sphygmomanometer.
Change in diastolic blood pressure. | Baseline and after 20 minutes of whole-body electrical stimulation.
  Safety will be assessed by monitoring diastolic blood pressure by sphygmomanometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No